CLINICAL TRIAL: NCT07077161
Title: Cabozantinib Dose Skipping as an Alternative to Dose Reductions
Acronym: SKIPPY 2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: dr. Tom van der Hulle (Other)
Responsible Party: Sponsor-Investigator, dr. Tom van der Hulle, Principal Investigator, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SKIPPY2; 2025-522962-58-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-08; First posted 2025-07-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Carcinoma (RCC)
Keywords: Renal Cell Carcinoma; RCC; Cabozantinib; pharmacokinetics
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: PK equivalence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard regimen (Active Comparator): taking 20mg or 40mg cabozantinib once daily with standard breakfast.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — For patients using 40mg the experimental regimen consists of 60mg once daily for 2 days followed by 1 skipping day (60-60-0 mg).
  For patients using 20mg the experimental regimen consists of 60mg once daily for 1 day followed by 2 skipping days (60-0-0 mg).
  In both cases cabozantinib is also taken with standard breakfast.

SUMMARY:
The goal of this study is to determine if an alternative cabozantinib dosing regimens results in a similar drug exposure compared to the standard regimens in patients with metastatic renal cell carcinoma (mRCC). All dosages of cabozantinib (20 ,40, 60mg) have the same price, and cabozantinib is eliminated very slowly by the body. This means that using fewer tablets could potentially lead to cost savings, while remaining equally effective.

The main questions it aims to answer are:

* Is the drug exposure from our experimental regimens similar to the standard dosing regimens?
* Do the experimental regimens affect the number of side effect and the patients' quality of life?

Participants will:

* Take cabozantinib according to either the experimental or standard dosage regimen for 4 weeks
* After 4 weeks: visit the clinic to collect some blood samples and complete two questionnaires.
* 1 and 3 days after this visit: visit the clinic to collect 1 blood sample.
* The day after the hospital visit: switch to the other dosing regimen and according to that regimen for another 4 weeks.
* After 4 weeks: visit the clinic to collect some blood samples and complete two questionnaires
* 1 and 3 days after this visit: visit the clinic to collect 1 blood sample.

DETAILED DESCRIPTION:
Standard regimens: 20 or 40mg once daily with standard breakfast

Experimental regimens:

* Instead of 20mg once daily: 60mg for one day, followed by two skipping days (60-0-0). Also taken with standard breakfast.
* Instead of 40mg once daily: 60mg for two days, followed by one skipping day (60-60-0). Also taken with standard breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent;
* Aged 18 years or older;
* Histologically confirmed advanced renal cell carcinoma;
* At least 4 weeks on a stable dosage of cabozantinib of 40 mg or 20 mg once daily as single-agent treatment or in combination with nivolumab;
* Acceptable tolerability and the need for dose reductions or treatment interruptions has been estimated as low;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* Estimated life expectancy of ≥6 months;
* No response evaluation planned during the study period.

Exclusion Criteria:

* Inability to follow the recommended standard breakfast;
* Gastrointestinal abnormalities influencing the absorption of cabozantinib, including active inflammatory bowel disease, malabsorption syndrome, and prior major surgery of the stomach, pancreas, liver or small bowel.
* Use of moderate or strong inhibitor of cytochrome P450 enzymes within 1 month of start of treatment with cabozantinib, including ketoconazole, grapefruit juice, clarithromycin, erythromycin, itraconazole and ritonavir.
* Use of moderate or strong inducer of cytochrome P450 enzymes within 1 month of start of treatment with cabozantinib, including rifampicin, phenytoin, carbamazepine, phenobarbital and herbal preparations containing St. John's Wort.
* Use of inhibitor of multidrug resistance-associated protein 2 within 1 month of start of treatment with cabozantinib, including cyclosporine, delavirdine, efavirenz, emtricitabine, benzbromarone and probenecid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the AUC0-72h of the experimental and the standard regimen. | From enrollment to the end of the study at approximately 2 months
  AUC is calculated by modeliing a PK curve from plasma concentrations. AUCs are compared between the standard and experimental regimen.
Comparison of blood trough concentration (Ctrough) | From enrollment to the end of the study at approximately 2 months
  Comparison of Ctrough, which is the plasma concentration of cabozantinib before ingestion of a dose cabozantinib, between the standard and experimental regimen.

SECONDARY OUTCOMES:
Health-economic cost-consequences | From enrollment to the end of the study at approximately 2 months
  Calculating the cost-savings of the alternative dosing regimens
Patients preference | From enrollment to the end of the study at 2 months
  Patients preference of one of the dosing regimens.
Quality of life score | From enrollment to the end of the study at approximately 2 months
  Fill in a questionnaires (EQ-5D-5L) about the quality of life. Which looks into two things:
  1. Five dimensions of health: mobility, self-care, daily activities, pain/disconfomrt and anxiety/some feelings. It uses a five point scale with 1 equally to no problem and 5 equally to extreme problems. It results in a score with 0 equally to dead and 1 equally to perfect health.
  2. Subjective assessment of one's own health on a scale from 0 to 100. Where 0 equals worst imaginable health and 100 equals best imaginable health.
Quality of life score | From enrollment to the end of the study at approximately 2 months
  Fill in a questionnaire (FKSI-19) with questions reflecting quality of life in patients with RCC. A question is answered using a 5-point scale where zero equals not at all and 4 equals very much. The higher the score the better the quality of life.
Side effects: nausea and/or diarrhea | From enrollment to the end of the study at approximately 2 months
  Total number of patients experiencing nausea and/or diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Tom van der Hulle, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- LUMC, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
To be determined in detail

REFERENCES:
- [Result] Tan Z, Voller S, Yin A, Rieborn A, Gelderblom AJ, van der Hulle T, Knibbe CAJ, Moes DJAR. Population Pharmacokinetics of Cabozantinib in Metastatic Renal Cell Carcinoma Patients: Towards Drug Expenses Saving Regimens. Clin Pharmacokinet. 2024 Jun;63(6):857-869. doi: 10.1007/s40262-024-01379-y. Epub 2024 Jun 14. PMID 38874883